CLINICAL TRIAL: NCT00878813
Title: Copeptin for Risk Stratification in Acute Stroke Patients: the CoRisk-study
Brief Title: Copeptin for Risk Stratification in Acute Stroke Patients: the CoRisk Study
Acronym: CoRisk
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Basel (Other); Charite University, Berlin, Germany (Other); Goethe University (Other)
Responsible Party: Sponsor
Other Study IDs: KEK 001/09
Record Dates: First submitted 2009-04-01; First posted 2009-04-09 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: Copeptin; Vasopressin; Stroke; Transient ischemic attack; Thrombolytic therapy; Prognosis; Complications
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Diabetes Insipidus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In all patients: 5 ml serum
  In patients undergoing intra-arterial revascularisation: 10 ml serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: All consecutive stroke patients undergoing acute intra-arterial revascularisation therapy
  Interventions: Procedure: Sampling of 15ml blood; Procedure: Blood-Sampling
- 2: All consecutive stroke patients undergoing acute intra-venous revascularisation therapy
  Interventions: Procedure: Sampling of 15ml blood; Procedure: Blood-Sampling
- 3: All consecutive stroke patients treated conservatively
  Interventions: Procedure: Sampling of 15ml blood
- 4: All consecutive TIA patients
  Interventions: Procedure: Sampling of 15ml blood

INTERVENTIONS:
Procedure: Sampling of 15ml blood — On admission, 2 x 7.5ml blood tubes will be drawn during the first routine blood sampling
Procedure: Blood-Sampling — On day 1 after intra-arterial thrombolysis, 2 x 7.5ml blood tubes on the following routine blood-sampling will be drawn.
  Groups: 1; 2

SUMMARY:
Prospective observational multicenter study to evaluate copeptin as a prognostic marker in patients with an acute cerebrovascular event. It includes four groups of patients, mainly depending on type of initial therapy (intra-arterial thrombolysis, intravenous thrombolysis, conservative treatment, TIA). The study takes place at the Emergency and neurological Department of the University of Bern, Switzerland; Department of Neurology, Goethe University of Frankfurt a.M. (Germany). Further participating centers are under discussion

DETAILED DESCRIPTION:
Background

The investigators in the Prolyse in Acute Cerebral Thromboembolism (PROACT) II study found that intra-arterial thrombolysis (IAT) with prourokinase within 6 hours after onset of symptoms was beneficial in patients with middle cerebral artery (MCA) occlusion. Intra-arterial thrombolysis (IAT) thus is an option for treatment of selected patients who have major stroke of <6 hours' duration due to occlusions of the MCA. Recently observational study showed that IAT was more beneficial than intra-venous thrombolysis (IVT) in the specific group of stroke patients presenting with hyperdense middle cerebral artery sign on CT, even though IAT was started later.

However complications after both reperfusion treatment modalities such as symptomatic intracerebral hemorrhage, malignant brain oedema, re-occlusion, infection, and seizures may occur. Unfortunately few clinical signs provide prognostic information for clear risk stratification. The guidelines for reperfusion therapies in Switzerland, Europe and the US do not include -for the time being- biomarkers in the decision-making-process. However there might be powerful biomarkers, which can serve as point of care tools for the risk stratification of candidates to receive thrombolysis. Plasma copeptin concentration has recently been shown to be an easy to determine, steady parameter which independently predicts functional outcome and death in patients with an acute ischemic stroke. Copeptin derives from a larger precursor peptide (pre-provasopressin) along with two other peptides, Vasopressin (AVP) and neurophysin II. Released in an equimolar ratio, the amount of copeptin mirrors the production of AVP. AVP plays an important role in the regulation of the hypothalamo-pituitary-adrenal (HPA) axis and, thus, reflecting the individual stress response. "Stressors" such as stroke are strong stimulators of the release of AVP. The close and reproducible relation of copeptin levels to the degree of activation of the stress axis is the basis of its usefulness as a biomarker. Early prognostic factors to predict mortality and outcome in stroke patients are important to guide and tailor early decision on treatment. In this context, copeptin may be helpful tool in the early risk stratification of stroke patients to guide the decision for reperfusion therapies.

Objective

To evaluate copeptin as prognostic tool to predict outcome in a well-defined cohort of stroke patients.

Methods

Step 1. All eligible patients in the emergency department or the neurological ward will be evaluated for enrollment into the study. On admission, 2 x 7.5ml- EDTA-blood tubes will be drawn during the first routine blood sampling, and 2 x 7.5ml-EDTA-blood tubes on the following routine blood-sampling. Copeptin levels will be assessed in a blinded batch analysis upon completion of the plasma asservation. Measurement will be performed with a new chemiluminescence sandwich immunoassay.

Step 2. All baseline data will be collected. CT or MRI will be performed 22 to 36 hours after IAT. All complications including death after the reperfusion therapies will be assessed until discharge.

Step 3. A telephone follow-up regarding morbidity and mortality will be obtained after 3 months. An unfavorable outcome will be defined as a mRs of 3 to 6

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients who are admitted to the emergency department with a clinical diagnosis of cerebrovascular event (TIA, stroke) within 24 hours of symptom onset

Exclusion Criteria:

Patients without informed consent. Patients discharged with a diagnosis different from stroke or TIA after diagnostic evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who are admitted to the emergency department of the Inselspital Bern - Switzerland with a clinical diagnosis of acute ischemic stroke within 24 hours of symptom onset. Inselspital Bern is a university based hospital with a catchment area of about 1.000.000 people
Sampling Method: Probability Sample
Enrollment: 1102 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Major disability or death | 90 days after qualifying event

SECONDARY OUTCOMES:
Symptomatic intracranial hemorrhage | until hospital discharge
Malignant brain oedema | until hospital discharge
Aspiration pneumonia | until hospital discharge
Seizure | until hospital discharge
Mortality | until hospital discharge
severe cerebrovascular re-event (i.e. new TIA, and stroke) | 90 days after qualifying event

CONTACTS AND LOCATIONS:
Overall Officials: Gian Marco De Marchis, MD, Principal Investigator — Inselspital, Bern University Hospital; Marcel Arnold, MD, Principal Investigator — Inselspital, Bern University Hospital; Mira Katan, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (4):
- Germany (2):
  - Abteilung für Neurologie Charité - Campus Benjamin Franklin, Berlin
  - Goethe University, Frankfurt am Main
- Switzerland (2):
  - Neurologische Klinik, Universitätsspital Basel, Basel
  - University Clinic for Neurology, Bern University Hospital, Bern

REFERENCES:
- [Background] Furlan A, Higashida R, Wechsler L, Gent M, Rowley H, Kase C, Pessin M, Ahuja A, Callahan F, Clark WM, Silver F, Rivera F. Intra-arterial prourokinase for acute ischemic stroke. The PROACT II study: a randomized controlled trial. Prolyse in Acute Cerebral Thromboembolism. JAMA. 1999 Dec 1;282(21):2003-11. doi: 10.1001/jama.282.21.2003. PMID 10591382
- [Background] Mattle HP, Arnold M, Georgiadis D, Baumann C, Nedeltchev K, Benninger D, Remonda L, von Budingen C, Diana A, Pangalu A, Schroth G, Baumgartner RW. Comparison of intraarterial and intravenous thrombolysis for ischemic stroke with hyperdense middle cerebral artery sign. Stroke. 2008 Feb;39(2):379-83. doi: 10.1161/STROKEAHA.107.492348. Epub 2007 Dec 20. PMID 18096842
- [Background] Maramattom BV, Bahn MM, Wijdicks EF. Which patient fares worse after early deterioration due to swelling from hemispheric stroke? Neurology. 2004 Dec 14;63(11):2142-5. doi: 10.1212/01.wnl.0000145626.30318.8a. PMID 15596765
- [Background] Aslanyan S, Weir CJ, Diener HC, Kaste M, Lees KR; GAIN International Steering Committee and Investigators. Pneumonia and urinary tract infection after acute ischaemic stroke: a tertiary analysis of the GAIN International trial. Eur J Neurol. 2004 Jan;11(1):49-53. doi: 10.1046/j.1468-1331.2003.00749.x. PMID 14692888
- [Background] Warach S, Latour LL. Evidence of reperfusion injury, exacerbated by thrombolytic therapy, in human focal brain ischemia using a novel imaging marker of early blood-brain barrier disruption. Stroke. 2004 Nov;35(11 Suppl 1):2659-61. doi: 10.1161/01.STR.0000144051.32131.09. Epub 2004 Oct 7. PMID 15472105
- [Background] Rubiera M, Alvarez-Sabin J, Ribo M, Montaner J, Santamarina E, Arenillas JF, Huertas R, Delgado P, Purroy F, Molina CA. Predictors of early arterial reocclusion after tissue plasminogen activator-induced recanalization in acute ischemic stroke. Stroke. 2005 Jul;36(7):1452-6. doi: 10.1161/01.STR.0000170711.43405.81. Epub 2005 Jun 9. PMID 15947260
- [Background] Adams HP Jr, del Zoppo G, Alberts MJ, Bhatt DL, Brass L, Furlan A, Grubb RL, Higashida RT, Jauch EC, Kidwell C, Lyden PD, Morgenstern LB, Qureshi AI, Rosenwasser RH, Scott PA, Wijdicks EF; American Heart Association; American Stroke Association Stroke Council; Clinical Cardiology Council; Cardiovascular Radiology and Intervention Council; Atherosclerotic Peripheral Vascular Disease and Quality of Care Outcomes in Research Interdisciplinary Working Groups. Guidelines for the early management of adults with ischemic stroke: a guideline from the American Heart Association/American Stroke Association Stroke Council, Clinical Cardiology Council, Cardiovascular Radiology and Intervention Council, and the Atherosclerotic Peripheral Vascular Disease and Quality of Care Outcomes in Research Interdisciplinary Working Groups: the American Academy of Neurology affirms the value of this guideline as an educational tool for neurologists. Stroke. 2007 May;38(5):1655-711. doi: 10.1161/STROKEAHA.107.181486. Epub 2007 Apr 12. PMID 17431204
- [Background] Toni D, Chamorro A, Kaste M, Lees K, Wahlgren NG, Hacke W; EUSI Executive Committee; EUSI Writing Committee. Acute treatment of ischaemic stroke. European Stroke Initiative. Cerebrovasc Dis. 2004;17 Suppl 2:30-46. doi: 10.1159/000074818. No abstract available. PMID 14707405
- [Background] Morgenthaler NG, Struck J, Alonso C, Bergmann A. Assay for the measurement of copeptin, a stable peptide derived from the precursor of vasopressin. Clin Chem. 2006 Jan;52(1):112-9. doi: 10.1373/clinchem.2005.060038. Epub 2005 Nov 3. PMID 16269513
- [Background] Katan M, Morgenthaler N, Widmer I, Puder JJ, Konig C, Muller B, Christ-Crain M. Copeptin, a stable peptide derived from the vasopressin precursor, correlates with the individual stress level. Neuro Endocrinol Lett. 2008 Jun;29(3):341-6. PMID 18580851
- [Derived] Rudin S, Kriemler L, Dittrich TD, Zietz A, Schweizer J, Arnold M, Peters N, Barinka F, Jung S, Arnold M, Fischer U, Rentsch K, Christ-Crain M, Katan M, De Marchis GM. Lipoprotein(a) as a blood marker for large artery atherosclerosis stroke etiology: validation in a prospective cohort from a swiss stroke center. Swiss Med Wkly. 2024 Apr 2;154:3633. doi: 10.57187/s.3633. PMID 38579294
- [Derived] De Marchis GM, Dankowski T, Konig IR, Fladt J, Fluri F, Gensicke H, Foerch C, Findling O, Kurmann R, Fischer U, Luft A, Buhl D, Engelter ST, Lyrer PA, Christ-Crain M, Arnold M, Katan M. A novel biomarker-based prognostic score in acute ischemic stroke: The CoRisk score. Neurology. 2019 Mar 26;92(13):e1517-e1525. doi: 10.1212/WNL.0000000000007177. Epub 2019 Mar 1. PMID 30824558
- [Derived] De Marchis GM, Weck A, Audebert H, Benik S, Foerch C, Buhl D, Schuetz P, Jung S, Seiler M, Morgenthaler NG, Mattle HP, Mueller B, Christ-Crain M, Arnold M, Katan M. Copeptin for the prediction of recurrent cerebrovascular events after transient ischemic attack: results from the CoRisk study. Stroke. 2014 Oct;45(10):2918-23. doi: 10.1161/STROKEAHA.114.005584. Epub 2014 Aug 28. PMID 25169950
- [Derived] De Marchis GM, Katan M, Weck A, Brekenfeld C, Mattle HP, Buhl D, Muller B, Christ-Crain M, Arnold M. Copeptin and risk stratification in patients with ischemic stroke and transient ischemic attack: the CoRisk study. Int J Stroke. 2013 Apr;8(3):214-8. doi: 10.1111/j.1747-4949.2011.00762.x. Epub 2012 Feb 15. PMID 22336226
- [Derived] Katan M, Elkind MS. Inflammatory and neuroendocrine biomarkers of prognosis after ischemic stroke. Expert Rev Neurother. 2011 Feb;11(2):225-39. doi: 10.1586/ern.10.200. PMID 21306210